CLINICAL TRIAL: NCT04498468
Title: Safety and Efficacy of Dexamethasone Ophthalmic Insert (Dextenza®) in the Management of Clinically Significant Dry Eye
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated prematurely due to administrative reasons; loss of several research personnel. Because of strict eligibility criteria, the investigators anticipated delays in completing enrollment and therefore decided to terminate early.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00246348
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dry Eye
Keywords: ocular surface disease; dexamethasone; ophthalmic steroids; keratoconjuntivitis sicca; dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Calcium Dobesilate; Punctal Plugs

STUDY DESIGN:
Intervention Model Description: Prospective, Double Masked, Interventional Study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the examining physician/outcomes accessor will be masked. The treating physician cannot be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Commercially available Sustained Release Dexamethasone, 0.4 mg intracannalicular insert (DEXTENZA® - Ocular Therapeutix, Bedford, MA)
  Interventions: Drug: Sustained Release Dexamethasone, 0.4 mg
- Control Arm (Sham Comparator): Commercially available EXTENDED WEAR SYNTHETIC ABSORBABLE PUNCTAL PLUG made of E-Caprolactone-L-Lactide copolymer (PCL) (Vera90™ - Elkridge, MD)
  Interventions: Other: E-Caprolactone-L-Lactide copolymer (PCL) punctal plug

INTERVENTIONS:
Drug: Sustained Release Dexamethasone, 0.4 mg — dexamethasone 0.4mg lacrimal insert
  Other Names: Dextenza
  Arms: Treatment Arm
Other: E-Caprolactone-L-Lactide copolymer (PCL) punctal plug — Control eye will receive a tear duct plug without the dexamethasone (EXTENDED WEAR SYNTHETIC ABSORBABLE PUNCTAL PLUG made of E-Caprolactone-L-Lactide copolymer (PCL). Absorbs in 60 to 180 days. Size 0.5mm which is comparable to the study treatment)
  Other Names: EXTENDED WEAR SYNTHETIC ABSORBABLE PUNCTAL PLUG
  Arms: Control Arm

SUMMARY:
To determine efficacy and safety profile of dexamethasone 0.4mg lacrimal insert in dry eye related ocular surface inflammation.

DETAILED DESCRIPTION:
Previous studies showed that dexamethasone and loteprednol topical drops have led to favorable results. However, the requirement of frequent instillation of drops by the patients is problematic causing discomfort and blurring of vision and requires remembering and dexterity for instillation, poor compliance is not uncommon. In addition Investigators believe that instillation of drops disturbs the homeostasis of the natural tear film due to physical and chemical trauma due to large drop volume (50 microliters) hammering on the eye surface (which can only hold 7 to 10 microliters). Particularly washing away of the mucin layer that holds all the "good ingredients" in the tears is harmful to the ocular surface. Therefore, "dropless" treatment of dry eye is desirable.

Dextenza® (dexamethasone ophthalmic insert, Ocular Therapeutix Inc., Bedford, MA) is a corticosteroid intracanalicular insert approved by US-FDA in November 2018 for the treatment of post-surgical ocular inflammation and pain. It is inserted into the lower lacrimal punctum and into the canaliculus. A single insert releases a 0.4 mg dose of dexamethasone for up to 30 days following insertion. Dextenza® is resorbable and does not require removal. Investigators hypothesize that Dextenza® could mimic short-term topical steroid use in a tapering manner in patients with clinically significant dry eye and show efficacy in improving its symptoms and signs, as was previously shown with other steroid preparations. If proven, the use of Dextenza® may shift paradigms in the management of the clinically significant ocular surface disease. To test this hypothesis, investigators propose to study the effects of Dextenza® in the treatment of clinically significant dry eye.

ELIGIBILITY:
Inclusion Criteria:

A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* Male or Female Age 18-100
* Capacity to give informed consent
* Ability to follow study direction and complete all study visits
* A previous or current diagnosis of dry eye by an eye care specialist, whereas treatment is requiring the use of a topical steroid
* Able to have a lacrimal plug placement into both lower puncta. If lower puncta are already plugged or cauterized/sealed, upper puncta will be used
* Females of childbearing potential unwilling to use reliable form(s) of birth control throughout study period
* Clinical diagnosis of dry eye syndrome (DES) or keratoconjunctivitis sicca (KCS), in which the following has been bilaterally documented in the ophthalmic and medical histories:

  i. history/diagnosis of dry eye ii. has taken or is on prescription drops (including but not limited to topical steroids, cyclosporine or lifitegrast)
* Presence of all of the following in both eyes at Baseline (Day 1):

  i. Total OSS of 3 or more with at least 2+ corneal staining (0-6) ii. Unanesthetized Schirmer level of <10 mm at 5 minutes iii. Presence of significant symptoms defined as 30mm or higher score of (1) eye dryness, or (2) eye fatigue, or (3) eye discomfort as measured using VAS, in both eyes. At the baseline visit, the most bothersome symptom (of the three) will be determined and used as the main symptom outcome measure throughout the study.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

* Use of Contact lenses within 1 week of screening visit or during the study
* Any ocular surgery (including tear duct cauterization) within the 3 months
* Inability to place a lacrimal device into upper or lower puncta of both eyes (if upper in R eye should be upper in the left eye and vice versa)
* Inability to participate in the wash out period
* Use of topical glaucoma medications (With exception of rescue medication)
* Pregnancy, nursing or intention of pregnancy or nursing in the study period.
* Monocular patients
* Uncontrolled systemic disease (defined as frequent or recent change in the medication regimen)
* Patients who are currently on with stable doses of oral steroids, topical cyclosporine or lifitigrast, topical tacrolimus or pimecrolimus are eligible as long as there has been no change in the dose in the last 3 months
* Patients who are on topical steroids (With exception of rescue medication) (Patients who have used steroids recently but have been off for at least 2 weeks will be eligible.)
* Current enrollment in any other investigational drug or device study or participation of study within 30 days of baseline visit.
* Known allergy or sensitivity to any of the clinical or experimental drugs used in this study including history of steroid response.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esen Akpek, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated information only will be shared with sponsor

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single-center, participant- and outcome assessor-masked, randomized controlled trial at the Ocular Surface Disease Clinic of Wilmer Eye Institute, The Johns Hopkins University School of Medicine in Baltimore, Maryland, USA.
Units Other Than Participants: eyes
Groups:
- All Study Participants: All participants received treatment and control.
  Treatment:
  Commercially available Sustained Release Dexamethasone, 0.4 mg intracannalicular insert (DEXTENZA® - Ocular Therapeutix, Bedford, MA) Sustained Release Dexamethasone, 0.4 mg: dexamethasone 0.4mg lacrimal insert
  Control:
  FCIProlong® made of E-Caprolactone-L-Lactide copolymer (PCL) (FCI Ophthalmics Inc., Pembroke, MA) E-Caprolactone-L-Lactide copolymer (PCL) punctal plug: Control eye will receive a tear duct plug without the dexamethasone (EXTENDED WEAR SYNTHETIC ABSORBABLE PUNCTAL PLUG made of E-Caprolactone-L-Lactide copolymer (PCL). Absorbs in 60 to 180 days. Size 0.5mm which is comparable to the study treatment)
Period: Overall Study
Arm/Group | All Study Participants
Started | 77; 154 eyes (Patients received both the treatment arm and the control arm - the eye that received the treatment was randomized. 77 participants, and thus 154 eyes, enrolled.)
Completed | 74; 148 eyes (2 patients were lost to follow-up. 1 patient did not complete their week 6 visit. All patients lost to follow-up were followed in PI's primary care post-study. Patients received both the treatment arm and the control arm - the eye that received the treatment was randomized. 74 participants, and thus 148 eyes, completed.)
Not Completed | 3; 6 eyes
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Only 75 (150 eyes) patients' data were analyzed at baseline as 2 patients were lost to follow-up before week 4.
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 75
Number analyzed (eyes) | 150
Age, Customized [Count of Participants; unit: Participants]
  Age Categories of Participants: 18-29 years | 2
  Age Categories of Participants: 30-39 years | 8
  Age Categories of Participants: 40-49 years | 10
  Age Categories of Participants: 50-59 years | 19
  Age Categories of Participants: 60-69 years | 23
  Age Categories of Participants: 70-79 years | 12
  Age Categories of Participants: 80 years or older | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 55
  More than one race | 0
  Unknown or Not Reported | 3
Posterior Blepharitis [Count of Participants; unit: Participants]
  Yes | 69
  No | 6
Visually Significant Cataract [Count of Participants; unit: Participants]
  Yes | 35
  No | 40
Anterior Blepharitis [Count of Participants; unit: Participants]
  Yes | 31
  No | 44
Punctal plugs [Count of Participants; unit: Participants]
  Yes | 27
  No | 48
Sjögren's [Count of Participants; unit: Participants]
  Yes | 27
  No | 48
Pseudophakia [Count of Participants; unit: Participants]
  Yes | 15
  No | 60
Conjunctival Scarring/Punctal stenosis [Count of Participants; unit: Participants]
  Yes | 6
  No | 69
Corneal Haze/Scarring [Count of Participants; unit: Participants]
  Yes | 3
  No | 72
Corneal Vascularization [Count of Participants; unit: Participants]
  Yes | 1
  No | 74
History of Corneal Ulceration [Count of Participants; unit: Participants]
  Yes | 2
  No | 73

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint as Assessed by Dry Eye Sign Using Ocular Surface Scale (OSS)
Description: OSS will be graded according to the Sjögren's International Collaborative Clinical Alliance (SICCA) grading system. Maximum possible fluorescein score (the punctate epithelial erosions grade + any extra points for modifiers [central staining, confluent staining, and filaments]) will be 6 and minimum of 0. Maximum possible conjunctival staining score (the punctate epithelial erosions grade on the temporal and nasal sides) will be 6 and minimum of 0. The total possible maximum OSS, derived by summing the corneal and conjunctival scores, will be 12 for each eye, and minimum OSS will be 0. Higher corneal, conjunctival, and staining scores represent worse outcomes.
  The difference between the average corneal staining in the treated arm versus the average corneal staining in the sham arm will be compared statistically.
Time Frame: 28 days
Population: Only 75 (150 eyes) patients' data were analyzed as 2 patients were lost to follow-up before 28 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Groups:
- Control Arm: FCIProlong® made of E-Caprolactone-L-Lactide copolymer (PCL) (FCI Ophthalmics Inc., Pembroke, MA)
  E-Caprolactone-L-Lactide copolymer (PCL) punctal plug: Control eye will receive a tear duct plug without the dexamethasone (EXTENDED WEAR SYNTHETIC ABSORBABLE PUNCTAL PLUG made of E-Caprolactone-L-Lactide copolymer (PCL). Absorbs in 60 to 180 days. Size 0.5mm which is comparable to the study treatment)
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 75 | 75
Number analyzed (eyes) | 75 | 75
score on a scale
  Day 28 Corneal Staining Mean Staining | 2.15 (1.31) | 2.70 (1.33)
  Day 28 Corneal Staining Mean Staining - Subgroup 18-59: number analyzed (Participants) | 39 | 39
  Day 28 Corneal Staining Mean Staining - Subgroup 18-59: number analyzed (eyes) | 39 | 39
  Day 28 Corneal Staining Mean Staining - Subgroup 18-59 | 2.14 (1.29) | 2.64 (1.55)
  Day 28 Corneal Staining Mean Staining - Subgroup 60+: number analyzed (Participants) | 36 | 36
  Day 28 Corneal Staining Mean Staining - Subgroup 60+: number analyzed (eyes) | 36 | 36
  Day 28 Corneal Staining Mean Staining - Subgroup 60+ | 2.13 (0.36) | 3.06 (1.12)
  Day 28 Corneal Staining Subgroup analysis by Sjögren's status - Yes: number analyzed (Participants) | 27 | 27
  Day 28 Corneal Staining Subgroup analysis by Sjögren's status - Yes: number analyzed (eyes) | 27 | 27
  Day 28 Corneal Staining Subgroup analysis by Sjögren's status - Yes | 2.54 (1.20) | 3.23 (1.42)
  Day 28 Corneal Staining Subgroup analysis by Sjögren's status - No: number analyzed (Participants) | 48 | 48
  Day 28 Corneal Staining Subgroup analysis by Sjögren's status - No: number analyzed (eyes) | 48 | 48
  Day 28 Corneal Staining Subgroup analysis by Sjögren's status - No | 1.82 (1.43) | 2.59 (1.23)
  Day 28 Conjunctival Staining Mean Staining | 3.01 (1.89) | 3.69 (1.69)
  Day 28 Conjunctival Staining Mean Staining - Subgroup 18-59: number analyzed (Participants) | 39 | 39
  Day 28 Conjunctival Staining Mean Staining - Subgroup 18-59: number analyzed (eyes) | 39 | 39
  Day 28 Conjunctival Staining Mean Staining - Subgroup 18-59 | 3.50 (2.35) | 2.69 (1.89)
  Day 28 Conjunctival Staining Mean Staining - Subgroup 60+: number analyzed (Participants) | 36 | 36
  Day 28 Conjunctival Staining Mean Staining - Subgroup 60+: number analyzed (eyes) | 36 | 36
  Day 28 Conjunctival Staining Mean Staining - Subgroup 60+ | 2.69 (1.89) | 3.88 (1.41)
  Day 28 Conjunctival Staining Subgroup analysis by Sjögren's status - Yes: number analyzed (Participants) | 27 | 27
  Day 28 Conjunctival Staining Subgroup analysis by Sjögren's status - Yes: number analyzed (eyes) | 27 | 27
  Day 28 Conjunctival Staining Subgroup analysis by Sjögren's status - Yes | 3.31 (2.39) | 4.09 (1.55)
  Day 28 Conjunctival Staining Subgroup analysis by Sjögren's status - No: number analyzed (Participants) | 48 | 48
  Day 28 Conjunctival Staining Subgroup analysis by Sjögren's status - No: number analyzed (eyes) | 48 | 48
  Day 28 Conjunctival Staining Subgroup analysis by Sjögren's status - No | 2.88 (1.93) | 3.59 (1.41)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Corneal staining analysis, day 28; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.91 to -0.19]
Statistical Analysis 2: Comparison: Treatment Arm vs Control Arm; Corneal staining sub-group analysis, day 28, 18-59 year old subgroup; Test type: Superiority; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.28 to 0.28]
Statistical Analysis 3: Comparison: Treatment Arm vs Control Arm; Corneal staining sub-group analysis, day 28, 60+ year old subgroup; Test type: Superiority; p = 0.047, t-test, 2 sided; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.86 to -0.02]
Statistical Analysis 4: Comparison: Treatment Arm vs Control Arm; Corneal staining sub-group analysis, day 28, Sjogren's subgroup; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.49 to 0.10]
Statistical Analysis 5: Comparison: Treatment Arm vs Control Arm; Corneal staining sub-group analysis, day 28, non-Sjogren's subgroup; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.67 to 0.14]
Statistical Analysis 6: Comparison: Treatment Arm vs Control Arm; Conjunctival staining analysis, day 28; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.05 to -0.30]
Statistical Analysis 7: Comparison: Treatment Arm vs Control Arm; Conjunctival staining sub-group analysis, day 28, 18-59 year old subgroup; Test type: Superiority; p = 0.58, t-test, 2 sided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.04 to 0.61]
Statistical Analysis 8: Comparison: Treatment Arm vs Control Arm; Conjunctival staining sub-group analysis, day 28, 60+ year old subgroup; Test type: Superiority; p = 0.021, t-test, 2 sided; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-2.17 to -0.21]
Statistical Analysis 9: Comparison: Treatment Arm vs Control Arm; Conjunctival staining sub-group analysis, day 28, Sjogren's subgroup; Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.88 to 0.34]
Statistical Analysis 10: Comparison: Treatment Arm vs Control Arm; Conjunctival staining sub-group analysis, day 28, non-Sjogren's subgroup; Test type: Superiority; p = 0.097, t-test, 2 sided; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.55 to 0.14]

2. Primary Outcome: Patient Reported Symptom
Description: (1)eye dryness, (2)eye discomfort, or (3)eye fatigue will be measured using visual analogue scale (0 to 100). The difference between the average bothersome symptom in the treated arm versus the average most bothersome symptom in the sham arm will be compared statistically. Higher VAS scores indicate worse eye dryness, discomfort, or fatigue.
Time Frame: 28 Days
Population: Only 75 (150 eyes) patients' data were analyzed as 2 patients were lost to follow-up before 28 days.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 75 | 75
Number analyzed (eyes) | 75 | 75
units on a scale
  Day 28 Eye Dryness VAS Mean Score | 49.3 (26.4) | 54.8 (23.0)
  Day 28 Eye Discomfort VAS Mean Score | 50.3 (27.7) | 50.6 (26.0)
  Day 28 Eye Fatigue VAS Mean Score | 43.7 (27.5) | 45.0 (26.7)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Eye dryness, day 28; Test type: Superiority; p = 0.069, t-test, 2 sided; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-11.4 to 0.4]
Statistical Analysis 2: Comparison: Treatment Arm vs Control Arm; VAS Eye discomfort, Day 28; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-7.0 to 6.3]
Statistical Analysis 3: Comparison: Treatment Arm vs Control Arm; VAS eye fatigue, day 28; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-5.8 to 3.1]

3. Secondary Outcome: Percentage of Subjects Achieving 2 Severity Grade Improvement in Corneal Staining
Description: Corneal staining responder analysis. Responder is defined as two full severity grade improvement in corneal staining. The percentage of subjects achieving two severity grades improvement in corneal staining (responders) in the treated arm versus sham arm will be compared statistically.
Time Frame: 42 days
Population: 74 (148 eyes) patients' data were analyzed as 3 patients were lost to follow-up before 42 days.
Measure: Number; unit: Percentage of responders
Units Other Than Participants: eyes
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 74 | 74
Number analyzed (eyes) | 74 | 74
Percentage of responders | 32 | 26
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Test type: Superiority; p = 0.42, McNemar; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.8 to 2.0]

4. Secondary Outcome: Percentage of Subjects Achieving Improvement in Their Most Bothersome Symptom
Description: Symptom responder analysis. Responder is defined as 30% or more improvement in the most bothersome symptom (VAS score is decreased by 30 points or more). The percentage of subjects achieving a 30% improvement in their most bothersome symptom (responders) in the treated arm versus the sham arm will be compared statistically.
Time Frame: 42 days
Population: 74 (148 eyes) patients' data were analyzed as 3 patients were lost to follow-up before 42 days.
Measure: Number; unit: Percentage of responders
Units Other Than Participants: eyes
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 74 | 74
Number analyzed (eyes) | 74 | 74
Percentage of responders | 38 | 37
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Test type: Superiority; p = 1.00, McNemar; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.76 to 1.42]

5. Other Pre Specified Outcome: Percentage of Participants With Intraocular Pressure Increase
Description: Intraocular Pressure (IOP) measurement obtained using applanation tonometry
Time Frame: At day 30 and day 42
Population: 75 (150 eyes) patients' data were analyzed at day 30. 74 (148 eyes) patients' data were analyzed at day 42.
Measure: Number; unit: percentage of subjects with IOP increase
Units Other Than Participants: eyes
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 75 | 75
Number analyzed (eyes) | 75 | 75
percentage of subjects with IOP increase
  Day 30 : Raised intraocular pressure (increase by 5-10 mm Hg from baseline) | 12 | 1
  Day 30 : Raised intraocular pressure (increase by >10 mm Hg from baseline) | 0 | 0
  Day 42 : Raised intraocular pressure (increase by 5-10 mm Hg from baseline): number analyzed (Participants) | 74 | 74
  Day 42 : Raised intraocular pressure (increase by 5-10 mm Hg from baseline): number analyzed (eyes) | 74 | 74
  Day 42 : Raised intraocular pressure (increase by 5-10 mm Hg from baseline) | 11 | 4
  Day 42 : Raised intraocular pressure (increase by >10 mm Hg from baseline): number analyzed (Participants) | 74 | 74
  Day 42 : Raised intraocular pressure (increase by >10 mm Hg from baseline): number analyzed (eyes) | 74 | 74
  Day 42 : Raised intraocular pressure (increase by >10 mm Hg from baseline) | 3 | 1

ADVERSE EVENTS:
Time Frame: Up to 42 days
Groups:
- Treatment Arm: Treatment:
  Commercially available Sustained Release Dexamethasone, 0.4 mg intracannalicular insert (DEXTENZA® - Ocular Therapeutix, Bedford, MA) Sustained Release Dexamethasone, 0.4 mg: dexamethasone 0.4mg lacrimal insert
- Control Arm: Control:
  FCIProlong® made of E-Caprolactone-L-Lactide copolymer (PCL) (FCI Ophthalmics Inc., Pembroke, MA) E-Caprolactone-L-Lactide copolymer (PCL) punctal plug: Control eye will receive a tear duct plug without the dexamethasone (EXTENDED WEAR SYNTHETIC ABSORBABLE PUNCTAL PLUG made of E-Caprolactone-L-Lactide copolymer (PCL). Absorbs in 60 to 180 days. Size 0.5mm which is comparable to the study treatment)
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/77 | 1/77
Other Adverse Events (participants affected / at risk) | 19/77 | 10/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=77) | Control Arm (N=77)
Day 14 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (77) — On 7/7/22, patient saw her neurosurgeon and was diagnosed with "high-grade glioma" and offered surgery, radiation, and chemotherapy. PI and pt. jointly decided to withdraw study consent in order for patient to focus on post neurosurgical recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=77) | Control Arm (N=77)
Week 6: Raised intraocular pressure (increase by 5-10 mm Hg from baseline) (Eye disorders) | 8 (8) | 3 (3)
Week 6: Raised intraocular pressure (increase by >10 mm Hg from baseline) (Eye disorders) | 2 (2) | 1 (1)
Week 6: Worsening of Corneal Fluorescein staining (increase by ≥2 from baseline) (Eye disorders) | 2 (2) | 2 (2)
Week 6: Worsening of conjunctival lissamine green staining (increase by ≥2 from baseline) (Eye disorders) | 7 (7) | 4 (4)

LIMITATIONS AND CAVEATS:
The study was not able to enroll its planned sample size. VAS, while consistently used in measuring clinical symptoms of illnesses, is limited in that patients may encounter difficulties in rating their symptomology, especially if the participants feel ambivalent towards the VAS prompts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04498468/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04498468/ICF_001.pdf